CLINICAL TRIAL: NCT06524960
Title: A Phase 1/2 Prospective, Randomized, Double-blind, Placebo-controlled Multi-center Clinical Trial to Determine the Safety and Efficacy of Denosumab in Improving Beta Cell Function and Glycemic Control Among Patients With Type 1 Diabetes
Brief Title: Denosumab for Type 1 Diabetes
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23797; JDRF Award:3-SRA-2023-1421-M-B (Other: JDRF)
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes, denosumab, HbA1c, beta cell function
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Subjects will be randomized to receive denosumab (Prolia) or normal saline placebo. Study treatment assignment will be blinded to study participants and investigators using a modified double-blind approach described below. The statistician at the primary site and the Research Pharmacist and Study Nurse administering denosumab (Prolia)/placebo at each site will know the treatment assignment and no disclosure of treatment will be allowed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Denosumab (Experimental): Denosumab 60 mg subcutaneous injection
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator): Normal Saline 1.0 ml subcutaneous injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Denosumab — Denosumab is a sterile, preservative-free, clear, colorless to pale yellow solution. Each 1 mL single-dose prefilled syringe of denosumab contains 60 mg denosumab (60 mg/mL solution), 4.7% sorbitol, 17 mM acetate, 0.01% polysorbate 20, Water for Injection (USP), and sodium hydroxide to a pH of 5.2.
  Arms: Denosumab
Other: Placebo — Placebo is 1 mL of normal saline drawn up in a commercially available syringe.
  Arms: Placebo

SUMMARY:
Type 1 diabetes (T1D) arises from abnormal immune cell-mediated injury to beta cells that make insulin. The injured beta cells can then no longer make the needed amount of insulin to stay healthy. However, in the early stages of T1D, some beta cells are still alive and functioning. Treatment to protect the beta cells against injury at this time could slow the progress of disease. Denosumab is an approved treatment for osteoporosis (a disease that thins and weakens the bones), high blood calcium levels, bone cancer, and other bone problems in patients who have cancer. The research team has found that the bone pathway that denosumab works on to treat these bone conditions also has effects on the health of the beta cells. Lab studies suggest that denosumab may protect and/or increase the number of beta cells and improve how well they work. This study will test whether denosumab is safe and improves beta cell function and blood sugar control in people with early T1D.

DETAILED DESCRIPTION:
This is a Phase 1/2, prospective, randomized, double-blind, placebo-controlled, multi-center clinical trial to evaluate the safety and efficacy of denosumab for improving beta cell function and glycemic control among patients with early T1D and detectable C-peptide. The efficacy of denosumab will be evaluated by changes in C-peptide level during mixed meal tolerance test and achieving a clinically meaningful HbA1c reduction at 12 months. Subjects will be followed for 12 months for adverse events and for changes in beta cell function and glycemic control parameters.

Subjects will be randomized with a 2:1 treatment to placebo ratio. The treatment group will enroll 30 subjects with the denosumab regimen of 60 mg given subcutaneously every 3 months for a total of 4 injections. The placebo arm will enroll 15 subjects and be administered with normal saline placebo given subcutaneously every 3 months for a total of 4 doses.

ELIGIBILITY:
Main Inclusion Criteria

* Age: Females 18-50 years; males 21-50 years (minimum age based on skeletal maturity)
* Diagnosis of type 1 diabetes (T1D) based on ADA Criteria:

  * Hyperglycemia (glycosylated hemoglobin (HbA1c) ≥ 6.5%; OR
  * fasting plasma glucose ≥ 126 mg/dl (7.0 mmol/L); OR
  * 2-hour plasma glucose ≥ 200 mg/dL (11.1 mmol/L) during an oral glucose tolerance test; OR
  * In a patient with classic symptoms of hyperglycemia or hyperglycemic crisis, a random plasma glucose ≥ 200 mg/dl (11.1 mmol/L)
* Documented history of at least one type 1 diabetes associated autoantibody

  * GAD specific autoantibodies (GADA);
  * Islet-antigen 2 specific autoantibody (IA-2A); and/or
  * Zinc Transporter 8 specific autoantibody (ZNT8A)
* Time from T1D diagnosis to screening MMTT must be ≥ 12 months but ≤ 5 years
* Non-fasting C-peptide concentrations of at least 0.2 nmol/L (0.6 ng/ml) at pre-screening and confirmed during a MMTT done at screening visit.
* Serum calcium (corrected for albumin)* within normal limits per site's local lab
* Agreement by women of childbearing potential (WOCBP) and males of childbearing potential to use a highly effective method of birth control for the course of the study through at least 5 months from the last dose of protocol therapy

Main Exclusion Criteria

* History of delayed puberty unless there is radiologic evidence of skeletal maturity
* Use of other investigational agents within 3 months of enrollment
* Vitamin D3 deficiency (< 30 ng/ml)
* History of anorexia and/or eating disorder
* BMI > 32 kg/m2
* HbA1c > 9.5%
* Severe hypoglycemia or diabetic ketoacidosis (DKA) within 3 months prior to screening. Subjects who had such episodes within 3-6 months prior to screening, must have written clearance from their treating physician.
* Use of any of the diabetes medications other than insulin within 3 months of enrollment (e.g., metformin, sulfonylurea, GLP-1 agonists, DPP4 inhibitors, Symlin, SGLT2-inhibitors, amylin)
* Treatment with any of the following drugs in past year: immunosuppressants, anticonvulsant therapy, adrenal or anabolic steroids, calcitonin, selective estrogen receptor modulator, sodium fluoride (other than dental treatment), teriparatide, abaloparatide, strontium or aromatase inhibitors; any history of bisphosphonate treatment.
* Bone fractures (excluding skull, facial bones, metacarpals, fingers, toes and spontaneous fractures associated with severe trauma) within the past 12 months
* Disorders associated with altered skeletal structure or function (Paget's disease, chronic liver disease (liver enzymes > twice the upper limit of normal), malignancy, hypoparathyroidism or hyperparathyroidism, acromegaly, Cushing's syndrome, hypopituitarism, chronic obstructive pulmonary disease, alcohol intake > 3 units/day)
* Significant dental/oral disease, including prior history or current evidence of osteonecrosis/osteomyelitis of the jaw, active dental or jaw condition requiring oral surgery, non-healed dental/oral surgery, or planned invasive dental procedures for the course of the study
* Pregnancy or actively breastfeeding (within 6 months prior to screening), or planning to become pregnant with 5 months after last dose of protocol therapy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2027-10-11 (Estimated); Study Completion 2027-10-11 (Estimated)

PRIMARY OUTCOMES:
Primary safety endpoint | up to 12 months
  To evaluate the safety of denosumab as assessed by the occurrence of adverse events (primary safety endpoint). Occurrence of treatment-related adverse events in denosumab group compared to placebo group during the 12 months.
  Toxicity: Toxicity and adverse events (except hypoglycemia and DKA) will be recorded in the eCRFs using the NCI CTCAE v 5.0 (See Section 7.0 for specific AEs). Hypoglycemia and DKA events will be defined per Section 14.1.1.
  - From treatment day through Month 12: All grade toxicities/AEs will be recorded.
  Safety will be assessed at baseline and at 3, 6, 9 and 12 months.
Primary efficacy endpoint | up to 12 months
  To evaluate the efficacy of denosumab in improving beta cell function in T1D subjects as measured by difference of mean area under the curve (AUC) of plasma C-peptide during 2-hr mixed meal tolerance test (MMTT) at baseline and 12 months after initiation of treatment (primary efficacy endpoint). Beta cell function as determined by the change in C-peptide AUC during MMTT in denosumab group will be compared to placebo group at 12 months from baseline.
  Change in Beta cell function (baseline and at 12 months)
  - Mixed meal tolerance test

SECONDARY OUTCOMES:
Beta cell function | Up to 6 months
  To evaluate the efficacy of denosumab in improving beta cell function as measured by C-peptide AUC during MMTT at 6 months. Beta cell function as determined by C-peptide AUC during MMTT in denosumab group will be compared to placebo group at 6 months.
  Beta cell function (baseline and at 6 months)
  - Mixed meal tolerance test
HbA1c improvement | up to 12 months
  To evaluate the efficacy of denosumab in improving HbA1c and insulin-dose adjusted HbA1c (IDAAIC) at 12 months. Changes in HbA1c and IDAAIC in denosumab group compared to placebo group.
  Glycemic Control (baseline and at 3, 6, 9 and 12 months)
  * HbA1c
  * IDAAIC is calculated as HbA1c (%) + [4 x insulin dose (units/kg/24hr)].

OTHER OUTCOMES:
Glucose variability | up to 12 months
  To evaluate the efficacy of denosumab on glucose variability as defined by time in target, and hypoglycemic and hyperglycemic ranges at 6 and 12 months. Glucose variability as defined by percent time in glycemic range (70-180 mg/dl and 70-140 mg/dl) and time spent in hypoglycemic and hyperglycemic ranges from continuous glucose monitoring data in denosumab group will be compared to placebo group.
  Glucose variability (baseline and at 6 and 12 months)
  - Continuous glucose monitoring
Insulin sensitivity | up to 12 months
  To evaluate the efficacy of denosumab on insulin sensitivity as calculated by the HOMA2 formula at 12 months. Insulin sensitivity as measured by HOMA2 in denosumab group will be compared to placebo group.
  Insulin sensitivity (baseline and at 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Fouad Kandeel, MD, PhD, Principal Investigator — City of Hope Medical Center; Rupangi Vasavada, PhD, Principal Investigator — City of Hope Medical Center
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - City of Hope Medical Center, Duarte, California
  - Indiana University, Indianapolis, Indiana